CLINICAL TRIAL: NCT00776841
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Escalating Single and Multiple-Dose Study of Aramchol in Healthy Male Volunteers
Brief Title: A Phase 1 Single and Multiple-Dose Study of Aramchol in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Medical Reserch (Industry)
Responsible Party: Dr. Itzchak Angel, Vice President, Research & Development, Galmed Medical Research
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROTOCOL No: TRC 037/10072
Record Dates: First submitted 2008-10-19; First posted 2008-10-21 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Phase-I; Hypercholesterolemia; Obesity; fatty liver; Part A: Healthy male volunteers Part B: Mildly overweight, otherwise healthy hypercholesterolemic male volunteers
MeSH Terms: conditions — Hypercholesterolemia; Obesity; Fatty Liver | interventions — aramchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Placebo (Placebo Comparator): Placebo control single dose
  Interventions: Drug: Aramchol
- Dose 1 (Experimental): Dose 30 mg
  Interventions: Drug: Aramchol
- Dose 2 (Experimental): Dose 100 mg
  Interventions: Drug: Aramchol
- Dose 3 (Experimental): Dose 300 mg
  Interventions: Drug: Aramchol
- Dose 4 (Experimental): Dose 900 mg
  Interventions: Drug: Aramchol
- Dose 1 repeated (Experimental): Dose 30 mg for 4 days
  Interventions: Drug: Aramchol
- Dose 2 repeated (Experimental): Dose high for 4 days
  Interventions: Drug: Aramchol

INTERVENTIONS:
Drug: Aramchol — 1.Aramchol in 16 healthy male subjects at single doses ranging between 30 and 900 mg (Part A) and in 30 overweight, mildly hypercholesterolemic, otherwise healthy male subjects receiving multiple doses (Part B)
  Other Names: 3β-arachidylamido-7α,12α,dihydroxy 5β-cholan-24-oic acid); fatty-acid bile-acid conjugate
Drug: Aramchol — Oral Aramchol at dose 30 mg to 900 mg
  Arms: Dose 1; Dose 2; Dose 3; Dose 4; Placebo
Drug: Aramchol — Oral Aramchol at doses 30 mg to 900 mg single dose and 30 mg and high dose for 4 days

SUMMARY:
A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Escalating Single and Multiple-Dose Study of Aramchol in Healthy Male Volunteers.

Primary Objectives:

1. To assess and characterize the safety and tolerability of Aramchol in 16 healthy male subjects at single doses ranging between 30 and 900 mg (Part A) and in 30 overweight, mildly hypercholesterolemic, otherwise healthy male subjects receiving multiple doses (Part B)
2. To assess the pharmacokinetics of Aramchol at the administered doses

DETAILED DESCRIPTION:
Number of Subjects:

Total: A total of 46 healthy subjects will be enrolled. Part A: Sixteen (16) subjects will participate in four, 8-person dosing periods. Each cohort will be alternately dosed twice.

Part B: Thirty (30) subjects will be enrolled in two, 15-person dose-ascending cohorts.

Main Inclusion Criteria:

Part A: Healthy male volunteers aged 18-50 (inclusive) years who have provided written informed consent Part B: Mildly overweight (25<BMI<33), with fasting cholesterol levels of 200-300 mg/% or LDL 100-180 mg/% and triglycerides < 200 mg/%, otherwise healthy male volunteers aged 18-50 (inclusive) years, who have provided written informed consent

ELIGIBILITY:
Inclusion Criteria:

* Part A: Healthy male volunteers aged 18-50 (inclusive) years who have provided written informed consent
* Part B: Mildly overweight (25<BMI <33), with fasting cholesterol levels of 200-300 mg/% or LDL 100-180 mg/% and triglycerides < 200 mg/%, otherwise healthy male volunteers aged 18-50 (inclusive) years, who have provided written informed consent

Major Exclusion Criteria:

* History of significant neurological (including history of seizures or EEG abnormalities), renal, cardiovascular (including known structural cardiac abnormalities or hypertension), respiratory (asthma), endocrinological, gastrointestinal, hematopoietic disease, neoplasm, psychological (marked anxiety, tension or agitation) or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medications.
* History of drug or alcohol abuse.
* Known allergy to any drug. Known allergy to any drug.
* Clinically significant abnormalities found in the screening physical exam.
* Significant abnormalities in clinical laboratory parameters (hematology, biochemistry, urinalysis) determined within 40 days of the start of the study and on Day (-1) before first dosing session. Parameters to be measured are those shown in Appendix 2.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability and Pharmacokinetics of Aramchol at single doses ranging between 30 and 900 mg (Part A) and in 30 overweight, mildly hypercholesterolemic, subjects receiving multiple doses (Part B) | day 1 to 6

SECONDARY OUTCOMES:
To assess and characterize the drug effect on lipid profile and functional pharmacodynamics following single and multiple dose administrations. | day 1 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, M.D., Principal Investigator — TASMC CLINICAL RESEARCH CENTER
Locations (1):
- Tasmc Clinical Research Center, Tel Aviv, Israel